CLINICAL TRIAL: NCT02592421
Title: Protocol 2: Elucidation of Mechanisms Responsible for the Increase in EGP Following SGLT2 Inhibition: Decrease in Plasma Glucose Conc or Change in Islet Hormone (Glucagon/Insulin) Secretion
Brief Title: SGLT2 Inhibition and Stimulation of Endogenous Glucose Production: Protocol 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20150668H; 5R01DK107680-02 (NIH)
Record Dates: First submitted 2015-10-14; First posted 2015-10-30 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Active Comparator): 20 subjects will receive dapagliflozin 10mg
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): 10 subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — SGLT2 inhibitor (dapagliflozin)
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
In Protocol 2, the investigators will determine the role of pancreatic hormones (increase in plasma glucagon and decrease in plasma insulin concentration) in the stimulation of EGP following SGLT2 inhibition.

DETAILED DESCRIPTION:
The inhibition of the renal (kidney) SGLT2 transporter has proven to be an effective therapeutic intervention to reduce plasma glucose levels (amount of glucose found in the liquid part of blood) and HbA1c.

In this study, the investigators hope to define the role of increased plasma glucagon, decline in plasma insulin, and fall in plasma glucose concentration. The investigators will examine whether the signal for the increase in EGP (endogenous glucose production) caused by glucosuria (an excess of sugar in the urine, typically associated with diabetes) is mediated via the decrease in plasma glucose and insulin concentrations, or by the increase in plasma glucagon concentration.

ELIGIBILITY:
Inclusion Criteria:

* T2DM subjects
* 18 - 70 yrs old
* BMI = 25-45 kg/m2
* Must be on a stable dose (more than 3 months) of monotherapy or combination therapy with metformin and/or a sulfonylurea
* HbA1c <10.0%
* Stable body weight (± 3 lbs) over preceding 3 months
* Do not participate in excessively heavy exercise

Exclusion Criteria:

* Subjects taking drugs known to affect glucose metabolism (other than metformin and sulfonylurea)
* Individuals with evidence of proliferative diabetic retinopathy, plasma creatinine >1.4 females or >1.5 males, or 24-hour urine albumin excretion > 300 mg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A. DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Alatrach M, Laichuthai N, Martinez R, Agyin C, Ali AM, Al-Jobori H, Lavynenko O, Adams J, Triplitt C, DeFronzo R, Cersosimo E, Abdul-Ghani M. Evidence Against an Important Role of Plasma Insulin and Glucagon Concentrations in the Increase in EGP Caused by SGLT2 Inhibitors. Diabetes. 2020 Apr;69(4):681-688. doi: 10.2337/db19-0770. Epub 2020 Jan 8. PMID 31915153

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg
  Dapagliflozin: SGLT2 inhibitor (dapagliflozin)
- Placebo: Subjects will receive placebo
  Placebo: Placebo Comparator
Period: Study 1
Arm/Group | Dapagliflozin | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0
Period: Study 2: Glucose Clamp Conditions
Arm/Group | Dapagliflozin | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0
Period: Study 3: Pancreatic Clamp Conditions
Arm/Group | Dapagliflozin | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (2) | 53 (2) | 53.5 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 4 | 16
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (0.7) | 31.4 (1.3) | 32 (2.85)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 6.9 (1.3) | 5.9 (1.5) | 6.4 (1.4)
Free Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 148 (8) | 127 (8) | 137 (8)
HBA1c (3 month blood glucose level measure) [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 7.5 (0.2) | 7.5 (0.1) | 7.5 (0.15)
Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min] | 97 (3) | 97 (3) | 97 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Glucose Concentration
Description: Change from baseline to the last hour of the study (240-300 minutes) in plasma glucose concentration
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
mg/dl
  Study 1 | -29.7 (3) | -17.2 (2.9)
  Study 2 with glucose clamp | 3.1 (0.9) | 0.9 (1.1)
  Study 3 with pancreatic clamp | -30.3 (3.5) | -2.3 (6.1)

2. Primary Outcome: Change in Endogenous Glucose Production (EGP)
Description: The change in endogenous glucose production is measured from baseline until the last hour of the study
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/kg.min
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
mg/kg.min
  Study 1 | 0.1 (0.1) | -0.56 (0.1)
  Study 2 with glucose clamp | -0.57 (0.12) | -1.28 (0.17)
  Study 3 with pancreatic clamp | -0.23 (0.09) | -0.48 (0.05)

3. Secondary Outcome: Change in Plasma Insulin During Measurement of EGP
Description: Measurement of change in plasma insulin concentration during measurement of of EGP from baseline to last hour of the study
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: microUnits/mL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
microUnits/mL
  Study 1 | 5 (1) | 3 (1)
  Study 2 with glucose clamp | 0 (1) | 0 (1)
  Study 3 with pancreatic clamp | 2 (1) | 0 (1)

4. Secondary Outcome: Change in Glucagon During EGP Measurement
Description: Measurement of change in glucagon during EGP measurement from baseline to the last hour of the study
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
ng/ml
  Study 1 | 5 (2) | -1 (2)
  Study 2 with glucose clamp | -6 (2) | -7 (3)
  Study 3 with pancreatic clamp | -1 (1) | -2 (2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study procedure, from baseline to 300 minutes
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 4/20 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=20) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) — Adverse event was experienced during study 3, the pancreatic clamp

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02592421/Prot_SAP_000.pdf